CLINICAL TRIAL: NCT04675112
Title: Genetically-informed Behavioral and Cognitive Interventions for the Management of Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gkouskou Kalliopi (Other)
Responsible Party: Sponsor-Investigator, Gkouskou Kalliopi, research associate, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No 208/2019
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A genetically informed intervention (Experimental): Group A patients are offered a genetically based approach to tinnitus management that includes a genetic test and at least three office based treatment sessions. A rationally-designed personalized management plan based on the genetic results is based on four single nucleotide polymorphisms (SNPs) of the dopamine and serotonin pathways, namely COMT rs4680, HTR2A rs7997012, HTR2A rs6311, and TPH2 rs4570625, that have been associated with behavioral or cognitive responses
  Interventions: Behavioral: Cognitive Behavioral Treatment (CBT) and Tinnitus Retraining Therapy (TRT)
- group B control (Other): In Group B, treatments are offered randomly taking care to offer CBT to equal number of patients as in Group A. In both groups, during the first visit, patients are offered a simple, few-minute tinnitus update and advice, relevant to their educational level and are being suggested that an average of 4 sessions are required over a period of approx. 4 months for making tinnitus noise less or not bothersome
  Interventions: Behavioral: Cognitive Behavioral Treatment (CBT) and Tinnitus Retraining Therapy (TRT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Treatment (CBT) and Tinnitus Retraining Therapy (TRT) — CBT is a psychologically informed treatment. Depending on individual patient needs, relevant areas of tinnitus education and management/self-management strategies, such as managing the emotional consequences of tinnitus, rapid relaxation, managing fear and avoidance behaviors and changing unhelpful thoughts and beliefs, are applied in accordance to a published manual [10].
  TRT is based on the neurophysiological model focusing more on education and sound therapy than on analytical cognitive and behavioral interventions. A TRT program is usually included in a management scheme with hearing aids.

SUMMARY:
Psychological and behavioral interventions, such as Cognitive Behavioral Treatment (CBT) and Tinnitus Retraining Therapy (TRT), are commonly applied either alone or in combination for the management of tinnitus but selection of the intervention model remains arbitrary. Our purpose is to evaluate the hypothesis that genetic markers may guide the choice of tinnitus treatment towards improved therapeutic outcomes. Patients with subjective idiopathic tinnitus are assigned to either a genetically-informed CBT or TRT intervention protocol based on the status of four single nucleotide polymorphisms (SNPs) of the dopamine and serotonin pathways, namely COMT rs4680, HTR2A rs7997012, HTR2A rs6311, and TPH2 rs4570625, that have been associated with behavioral or cognitive responses (Group A), or to a conventional approach (Group B) in which the choice of treatment was not directed by genotypic data. Tinnitus Handicap Index (THI) scores of perceived tinnitus severity are recorded at the initial and at the fourth session of treatment using appropriate questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with bothersome bilateral non-pulsative tinnitus and hearing loss

Exclusion Criteria:

* no major comorbidities
* no psychiatric history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | 4 months
  Upon a detailed history and an integrated ENT and audiological examination, the patients are asked to answer the THI twice (pre and post treatment), a questionnaire that quantifies the impact of tinnitus on everyday function. It is psychometrically robust and demonstrates adequate reliability and validity [9]

CONTACTS AND LOCATIONS:
Locations (1):
- ENT clinic, Athens, Greece

IPD SHARING:
Plan to Share IPD: No